CLINICAL TRIAL: NCT04368897
Title: In-vitro Diagnostic Test to Predict COVID-19 Mortality and Disease Severity
Status: Withdrawn | Type: Observational
Why Stopped: Not able to recruit subjects
Sponsor: Applied Biology, Inc. (Industry)
Collaborators: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Other Study IDs: AB-IVD-CoV-001
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2022-02

CONDITIONS: SARS-CoV 2; COVID; COVID-19; Androgenetic Alopecia; Androgen Receptor Abnormal; Androgen Deficiency
MeSH Terms: conditions — COVID-19; Alopecia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva DNA sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Male Patients: Males with laboratory confirmed SARS-CoV-2 infection
  Interventions: Diagnostic Test: CAG length <22; Diagnostic Test: CAG length >=22

INTERVENTIONS:
Diagnostic Test: CAG length <22 — CAG repeat length in exon 1 of AR gene
  Other Names: Genetic Test - Short CAG Allele
Diagnostic Test: CAG length >=22 — CAG repeat length in exon 1 of AR gene
  Other Names: Genetic Test - Long CAG Allele

SUMMARY:
The COVID-19 Androgen Sensitivity Test is a non-invasive In-Vitro Diagnostic device that utilizes Next Generation Sequencing Technology (NGS). The results of the test are used by a physician to assess the risk of developing severe symptoms following COVID-19 infection, The COVID-19 Androgen Sensitivity Test requires a health care professional to collect a DNA sample using an FDA cleared DNA sample collection kit.

DETAILED DESCRIPTION:
In late 2019, a novel coronavirus, subsequently named SARS-CoV-2 (COVID-19), was first reported in Hubei province in China. Since it was first reported, a worldwide pandemic has ensued affecting more than 450,000 individuals as of March 2020. In the midst of the pandemic, epidemiological reports unveiled a disproportionate low rate of severe cases among adult females compared to adult males, 42% and 58%, respectively. Similarly, the rate of severe cases among pre-pubescent children was exceptionally low at 0.6%. An explanation for the skewed prevalence of severe COVID-19 infection in adult males has yet to be elucidated.

In newborns, it has long been recognized that male infants are more susceptible to respiratory distress syndrome and less likely to respond to prenatal glucocorticoid therapy to protect against respiratory distress. Respiratory distress is intimately tied to the production of pulmonary surfactant, e.g., pulmonary surfactant proteins have been demonstrated to protect against influenza A. In animal studies, it was demonstrated that a sexual dimorphism in fetal pulmonary surfactant production is influenced by the androgen receptor (AR). For example, in rabbits, dihydrotestosterone was shown to inhibit fetal pulmonary surfactant production in both males and females while an anti-androgen, flutamide, was demonstrated to remove the sexual dimorphism in surfactant production. While severe COVID-19 symptoms are primarily manifested in older adults, the similar sexual dimorphism in the severity of respiratory disease is of interest. In addition, AR expression is low prior to pubertal maturation and may contribute to the low incidence of severe COVID-19 infection in children. As such, the investigators propose that the lower rate of severe COVID-19 infection in female patients may be attributed to lower androgen receptor expression.

Additional evidence to the possible implication of androgens in COVID-19 infection severity is found in the molecular mechanism required for SARS-CoV-2 infectivity. SARS-CoV-2 is part of the coronavirus family of viruses including SARS-CoV-1 and MERS-CoV. Coronavirus predominantly infects type II pneumocytes in the human lung. Previously, it was demonstrated that SARS-CoV-2 cell entry depends on priming of a viral spike surface protein by transmembrane protease serine 2 (TMPRSS2) present in the host. In type II pneumocytes, TMPRSS2 expression is associated with an increase in androgen receptor (AR) expression, specifically connecting AR expression to SARS-CoV-2, due to AR-regulated TMPRSS2 gene promoter. Moreover, angiotensin converting enzyme 2 (ACE2) has been recognized as the attachment molecule to the viral spike surface protein, thus termed the "receptor of SARS-CoV-2". Interestingly, ACE2 has been shown to have reduced activity by the decrease of androgen hormones (experimental orchidectomy), possibly by decreased expression of ACE2.

A well known polymorphism of the androgen receptor is a CAG repeat in the first exon of AR gene. The number of CAG repeats has been correlated with AR function and expression. The primary purpose of this study is to evaluate the association of AR gene polymorphisms with disease severity and mortality following COVID-19 infection. If an association can be elucidated, it would imply novel treatment modalities. For example, the activation of AR can be reduced by several classes of drugs including androgen receptor antagonists, androgen synthesis inhibitors and antigonadotropins.

ELIGIBILITY:
Inclusion Criteria:

* Male over the age of 18
* First time present at the site
* Laboratory confirmed SARS-CoV-2 infection
* Able to give informed consent

Exclusion Criteria:

* Unable to give informed consent
* Diagnosed with an additional respiratory co-infection
* XXY males

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Self description
Study Population: Patients admitted to the hospital due to COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Hospital-free days to Day 28 [ Time Frame: 28 days] | 28 days
  Defined as 28 days minus the number of days from randomization to discharge home. If a patient has not been discharged home prior to day 28 or dies prior to day 28, hospital free days will be zero.
1. Severity of Disease | Day 28
  Defined as discharged, hospitalization, admission to intensive care unit [ICU] and death

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Herrera, MD, Principal Investigator — Hospital Universitario Ramon y Cajal; Carlos Wambier, MD, Study Director — Brown University
Locations (1):
- Hospital Universitario Ramon y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goren A, McCoy J, Wambier CG, Vano-Galvan S, Shapiro J, Dhurat R, Washenik K, Lotti T. What does androgenetic alopecia have to do with COVID-19? An insight into a potential new therapy. Dermatol Ther. 2020 Jul;33(4):e13365. doi: 10.1111/dth.13365. Epub 2020 Apr 8. No abstract available. PMID 32237190
- [Result] Wambier CG, Goren A. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection is likely to be androgen mediated. J Am Acad Dermatol. 2020 Jul;83(1):308-309. doi: 10.1016/j.jaad.2020.04.032. Epub 2020 Apr 10. PMID 32283245
- [Result] Goren A, Vano-Galvan S, Wambier CG, McCoy J, Gomez-Zubiaur A, Moreno-Arrones OM, Shapiro J, Sinclair RD, Gold MH, Kovacevic M, Mesinkovska NA, Goldust M, Washenik K. A preliminary observation: Male pattern hair loss among hospitalized COVID-19 patients in Spain - A potential clue to the role of androgens in COVID-19 severity. J Cosmet Dermatol. 2020 Jul;19(7):1545-1547. doi: 10.1111/jocd.13443. Epub 2020 Apr 23. PMID 32301221
- [Result] McCoy J, Wambier CG, Vano-Galvan S, Shapiro J, Sinclair R, Ramos PM, Washenik K, Andrade M, Herrera S, Goren A. Racial variations in COVID-19 deaths may be due to androgen receptor genetic variants associated with prostate cancer and androgenetic alopecia. Are anti-androgens a potential treatment for COVID-19? J Cosmet Dermatol. 2020 Jul;19(7):1542-1543. doi: 10.1111/jocd.13455. Epub 2020 Jun 14. No abstract available. PMID 32333494